CLINICAL TRIAL: NCT02006836
Title: Glycemic Index & Glycemic Responses to Majia Pomelos
Brief Title: Glycemic Responses to Majia Pomelos in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xuefeng Yu, Director of Division of Endocrinology, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Tongji201201
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes
Keywords: glycemic index; glycemic response; diabetes; pomelo
MeSH Terms: conditions — Diabetes Mellitus | interventions — Glucose; Insulin; Insulin Aspart; Proto-Oncogene Proteins c-met; Diet; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Diabetic (Other): Diabetic patients use metformin or only on diet control(met or diet).18 of the patients were on metformin treatment and 2 patients were on diet control due to the early stage of this disease. On the first test day we utilized 50 g of glucose dissolved in 200 ml water. The second day was washout day. On the third day we used 922 g of Majia pomelos which contained 50 g carbohydrate.This group of diabetic patients enrolled for the case control period.
  Interventions: Dietary Supplement: Pomelo; Dietary Supplement: Glucose; Drug: met or diet
- Healthy (Other): On the first test day we utilized 50 g of glucose dissolved in 200 ml water. The second day was washout day. On the third day we used 922 g of Majia pomelos which contained 50 g carbohydrate.This group of volunteers enrolled for the case control period.
  Interventions: Dietary Supplement: Pomelo; Dietary Supplement: Glucose
- Diabetic 2 - without pomelo (Other): Patients of Diabetic 2 group were on CSII treatment with insulin subcutaneous pump.The scheme and dose of CSII for each patients were adjusted on the first 3 test days to optimize glucose control, followed by 3-day CSII treatment without change of insulin dose. On the 7th test day, patients consumed 100g Majia pomelos after meals (breakfast, lunch and dinner) for 3 test days. This arm refers to the group on the 4th to 6th day with a constant dose of insulin and did not consumed Majia pomelos after meals, and this intervention was defined as blank.
  Interventions: Other: Blank; Drug: Insulin
- Diabetic 2 - with pomelo (Other): Patients of Diabetic 2 group were on CSII treatment with insulin subcutaneous pump.The scheme and dose of CSII for each patients were adjusted on the first 3 test days to optimize glucose control, followed by 3-day CSII treatment without change of insulin dose. On the 7th test day, patients consumed 100g Majia pomelos after meals (breakfast, lunch and dinner) for 3 test days. This arm refers to the group on the 7th to 9th day with a constant dose of insulin and consumed 100g Majia pomelos after meals (breakfast, lunch and dinner).
  Interventions: Dietary Supplement: Pomelo; Drug: Insulin

INTERVENTIONS:
Dietary Supplement: Pomelo — The sugar content of the pomelo was 5.86% of full weight, and we use 922g Majia pomelos which contained about 50g sugar equal to 50g glucose for GI measurement.
  Other Names: Majia pomelos; Citrus grandis cv. Majiayou
  Arms: Diabetic; Diabetic 2 - with pomelo; Healthy
Dietary Supplement: Glucose — We dissolved 50 g of glucose in 200 ml water.
  Other Names: Anhydrous glucose
  Arms: Diabetic; Healthy
Other: Blank — For the self-control period the diabetic patients underwent 3-day CSII treatment without change of insulin dose and we did not applied any intervention.
  Arms: Diabetic 2 - without pomelo
Drug: Insulin — Patients who were included in the test of glycemic responses to postprandial pomelo consumption were hospitalized with the treatment of Continuous Subcutaneous Insulin Infusion(CSII), and the insulin for CSII was insulin aspart(NovoRapid).
  Other Names: Insulin aspart; NovoRapid
  Arms: Diabetic 2 - with pomelo; Diabetic 2 - without pomelo
Drug: met or diet — In diabetic group, 20 diabetic patients were included for GI measurement , 18 of whom were on metformin treatment. Only 2 patients were on diet control due to the early stage of this disease.
  Other Names: metformin; diet control
  Arms: Diabetic

SUMMARY:
Food intake has a great influence on blood glucose of patients with diabetes. This study was designed to determine the glycemic index (GI) of a particular pomelo named Majia pomelo and its effects on postprandial glucose (PPG) excursions in both healthy subjects and patients with type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the GI and effects on glucose excursion of Majia pomelo in both healthy and diabetic subjects. The results may help diabetic subjects and their health care providers in developing a diet that is both medically and culturally appropriate.

ELIGIBILITY:
Inclusion Criteria:

* In the diabetic and diabetic 2 groups, it required that their diabetes was controlled (HbA1c ≤ 8%) on diet with or without metformin.

Exclusion Criteria:

* Morbid obesity (BMI > 40 kg/m2)
* Pre diabetes
* Pregnancy
* Presence of gastroenterological disorders
* Alimentary tract surgery
* A history of gastroenteritis in the prior six months
* Any alcohol intake
* Smoking
* Taking any medications (except metformin)
* Poorly controlled diabetes (HbA1c > 8%)
* Presence of chronic diseases (such as bronchial asthma or rheumatoid arthritis) or acute illness (such as upper respiratory tract or urinary tract infection)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng Yu, PhD MD, Principal Investigator — Division of Endocrinology, Tongji Hospital, Huazhong University of Science & Technology
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period : 2013.1-2013.12, and there are two periods of the study. Case-control period: month 1- month 6, self-control period: month 7-month 12.
  Study participants were recruited from Tongji Hospital and local poster advertisements
Pre-assignment Details: In diabetic group, patients had taken metformin or pioglitazone or only on life modification for at least 3 months. In diabetic 2 group, patients were hospitalized treated with insulin for at least 6 days.We matched each of the diabetic patients to a healthy control according to age, BMI, and gender in the case-control period.
Groups:
- Case-Control: Diabetic; Case-Control: Healthy: For case-control period and for GI measurement. 50 g of glucose dissolved in 200 ml water followed sequentially by 50g carbohydrate equivalents of 922g Majia pomelos.
- Self-Control: Diabetic 2: For self-control period. Patients of Diabetic 2 group were on CSII treatment with insulin subcutaneous pump.The scheme and dose of CSII for each patients were adjusted on the first 3 test days to optimize glucose control, followed by 3-day CSII treatment without change of insulin dose. On the 7th test day, patients consumed 100g Majia pomelos after meals (breakfast, lunch and dinner) for 3 test days.
  On the 4th to 6th day, patients with a constant dose of insulin did not consume Majia pomelos after meals, and this intervention was defined as blank.
  On the 7th to 9th day, patients with the same dose of insulin consumed 100g Majia pomelos after meals (breakfast, lunch and dinner).
Period: Case-control Period: Month 1- Month 6
Arm/Group | Case-Control: Diabetic | Case-Control: Healthy | Self-Control: Diabetic 2
Started | 20 | 20 | 0
Completed | 20 | 20 | 0
Not Completed | 0 | 0 | 0
Period: Self-control Period: Month 7-month 12
Arm/Group | Case-Control: Diabetic | Case-Control: Healthy | Self-Control: Diabetic 2
Started | 0 | 0 | 19
Completed | 0 | 0 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We chose the petients who met the inclusion/exclusion criteria and completed the study for the final analysis.
Groups:
- Diabetic; Healthy: For case-control period and for GI measurement. 50 g of glucose dissolved in 200 ml water followed sequentially by 50g carbohydrate equivalents of 922g Majia pomelos.
- Diabetic 2: For self-control period. The scheme and dose of Continuous Subcutaneous Insulin Infusion (CSII) for each patients were adjusted on the first 3 test days to optimize glucose control, followed by 3-day CSII treatment without change of insulin dose. On the 7th test day, patients consumed 100g Majia pomelos after meals (breakfast, lunch and dinner) for 3 test days.
- Total: Total of all reporting groups
Arm/Group | Diabetic | Healthy | Diabetic 2 | Total
Number analyzed (Participants) | 20 | 20 | 19 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.15 (2.52) | 54.30 (2.42) | 50.42 (2.48) | 53.34 (1.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 23
  Male | 12 | 12 | 12 | 36
Region of Enrollment [Number; unit: participants]
  China | 20 | 20 | 19 | 59
Body weight [Mean (Standard Deviation); unit: kg] | 69 (2.9) | 66.24 (2.43) | 68.59 (2.64) | 67.93 (1.52)
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.51 (0.97) | 24.49 (0.64) | 24.76 (0.69) | 24.92 (0.45)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 129.8 (3.5) | 124.65 (3.66) | 128.32 (3.36) | 127.58 (2.01)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 78.05 (2.11) | 75.25 (1.96) | 82.0 (1.74) | 78.37 (1.16)
HbA1c [Mean (Standard Deviation); unit: %] | 7.53 (0.45) | 5.57 (0.06) | 10.06 (0.61) | 7.60 (0.33)

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Index
Description: Glycemic index (GI) measurement was carried out after an overnight fast on 2 occasions in every subject, each test being separated from the next by a "washout" day.The first test day utilized 50 g of glucose dissolved in 200 ml water followed sequentially by 50g carbohydrate equivalents of the Majia pomelos. Venous blood samples were collected and monitored during 3 hrs for both the healthy and T2DM individuals at 0, 30, 60, 90, 120, 150, and 180 min. Areas under the curves (AUC) of blood glucose concentrations were obtained. The 50 g of glucose was used as the reference (GI = 100) according to the literature. The AUC under the incremental glycemic-response curves for Majia were expressed as a percentage of the areas under the glucose curves for the same subject. The resulting values for all subjects were averaged to calculate the GI.
  GI measurement is only calculated in case-control period.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: percentage of AUC from GI100
Groups:
- Diabetic; Healthy: For case-control period. 50 g of glucose dissolved in 200 ml water followed sequentially by 50g carbohydrate equivalents of 922g Majia pomelos.
Arm/Group | Diabetic | Healthy
Number analyzed (Participants) | 20 | 20
percentage of AUC from GI100 | 76.79 (1.83) | 86.92 (2.17)
Statistical Analysis 1: Comparison: Diabetic vs Healthy; H0: GI of pomelo for diabetic patients - GI of pomelo for healthy people = 0 H1: GI of pomelo for diabetic patients - GI of pomelo for healthy people > 0 α=5%; Test type: Superiority or Other; p = 0.005, t-test, 1 sided

2. Primary Outcome: ∆g of Breakfast With/Without Pomelo
Description: After the dose of CSII for each patients were adjusted on the first 3 test days to optimize glucose control, there were 3-day CSII treatment without change of insulin dose. Capillary blood samples were detected before and after meals. Glucose difference (∆g) before and after breakfast were obtained and analyzed.
  * g of breasfast without pomelo=mean of 3 days of postprandial blood glucose after breakfast - mean of 3 days of blood glucose before this breakfast.
  * g of breasfast with pomelo=mean of 3 days of postprandial blood glucose after breakfast - mean of 3 days of blood glucose before this breakfast.
Time Frame: 9 days
Population: The patients met the inclusion/exclusion criteria and completed the study.
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Diabetic 2 - Without Pomelo | Diabetic 2 - With Pomelo
Number analyzed (Participants) | 19 | 19
mmol/l | 2.93 (0.72) | 3.61 (0.58)
Statistical Analysis 1: Comparison: Diabetic 2 - Without Pomelo vs Diabetic 2 - With Pomelo; H0：∆g after breakfast- ∆g before breakfast = 0 H1：∆g after breakfast- ∆g before breakfast > 0 α=5% * g of breasfast without pomelo=mean of 3 days of postprandial blood glucose after breakfast - mean of 3 days of blood glucose before this breakfast. * g of breasfast with pomelo=mean of 3 days of postprandial blood glucose after breakfast - mean of 3 days of blood glucose before this breakfast; Test type: Superiority or Other; p > 0.05, t-test, 1 sided

3. Primary Outcome: ∆g of Lunch With/Without Pomelo
Description: After the dose of CSII for each patients were adjusted on the first 3 test days to optimize glucose control, there were 3-day CSII treatment without change of insulin dose. Capillary blood samples were detected before and after meals. Glucose difference (∆g) before and after lunch were obtained and analyzed.
  * g of lunch without pomelo=mean of 3 days of postprandial blood glucose after lunch without pomelo - mean of 3 days of blood glucose before this lunch.
  * g of lunch with pomelo=mean of 3 days of postprandial blood glucose after lunch with pomelo- mean of 3 days of blood glucose before this lunch.
Time Frame: 9 days
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Diabetic 2 - Without Pomelo | Diabetic 2 - With Pomelo
Number analyzed (Participants) | 19 | 19
mmol/l | 1.39 (0.63) | 2.87 (0.47)
Statistical Analysis 1: Comparison: Diabetic 2 - Without Pomelo vs Diabetic 2 - With Pomelo; H0：∆g after lunch - ∆g before lunch = 0 H1：∆g after lunch - ∆g before lunch > 0 α=5% * g of lunch without pomelo=mean of 3 days of postprandial blood glucose after lunch - mean of 3 days of blood glucose before this lunch. * g of lunch with pomelo=mean of 3 days of postprandial blood glucose after lunch - mean of 3 days of blood glucose before this lunch; Test type: Superiority or Other; p > 0.05, t-test, 1 sided

4. Primary Outcome: ∆g of Dinner With/Without Pomelo
Description: After the dose of CSII for each patients were adjusted on the first 3 test days to optimize glucose control, there were 3-day CSII treatment without change of insulin dose. Capillary blood samples were detected before and after meals. Glucose difference (∆g) before and after dinner were obtained and analyzed.
  * g of dinner without pomelo=mean of 3 days of postprandial blood glucose after dinner without pomelo - mean of 3 days of blood glucose before this dinner.
  * g of dinner with pomelo=mean of 3 days of postprandial blood glucose after dinner with pomelo - mean of 3 days of blood glucose before this dinner.
Time Frame: 9 days
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Diabetic 2 - Without Pomelo | Diabetic 2 - With Pomelo
Number analyzed (Participants) | 19 | 19
mmol/l | 0.34 (0.41) | 1.41 (0.24)
Statistical Analysis 1: Comparison: Diabetic 2 - Without Pomelo vs Diabetic 2 - With Pomelo; H0：∆g after dinner- ∆g before dinner = 0 H1：∆g after dinner- ∆g before dinner > 0 α=5% * g of dinner without pomelo=mean of 3 days of postprandial blood glucose after dinner - mean of 3 days of blood glucose before this dinner. * g of dinner with pomelo=mean of 3 days of postprandial blood glucose after dinner - mean of 3 days of blood glucose before this dinner; Test type: Superiority or Other; p > 0.05, t-test, 1 sided

5. Primary Outcome: AUCs With/Without Pomelo
Description: Patients of Diabetic 2 group were on CSII treatment with insulin subcutaneous pump.The scheme and dose of CSII for each patients were adjusted on the first 3 test days to optimize glucose control, followed by 3-day CSII treatment without change of insulin dose. On the 7th test day, patients consumed 100g Majia pomelos after meals (breakfast, lunch and dinner) for 3 test days. Capillary blood samples were detected before and after meals, 10pm, and 3am. Mean of each time point(before breakfast, 2 hours after breakfast, before lunch, 2 hours after lunch, before dinner, 2 hours after dinner,10pm, and 3am ) of blood glucose concentrations on 4th to 6th day（without pomelo） were calculated and so as each time point of blood glucose concentrations on 7th to 9th day (with pomelo). Areas under the curves (AUC) of mean blood glucose concentrations of each time point were obtained with/without pomelo.
Time Frame: 9 days
Measure: Mean (Standard Deviation); unit: mmol*hour/L
Arm/Group | Diabetic 2 - Without Pomelo | Diabetic 2 - With Pomelo
Number analyzed (Participants) | 19 | 19
mmol*hour/L | 164.04 (7.58) | 163.07 (6.90)
Statistical Analysis 1: Comparison: Diabetic 2 - Without Pomelo vs Diabetic 2 - With Pomelo; H0: AUC; Test type: Superiority or Other; p > 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 3 days for Diabetic and Healthy group. 9 days for Diabetic 2 - without pomelo and Diabetic 2 - with pomelo group.
Groups:
- Diabetic: Diabetic patients use oral antidiabetic drugs(metformin or pioglitazone or both) or only life style modification. On the first test day we utilized 50 g of glucose dissolved in 200 ml water. The second day was washout day. On the third day we used 922 g of Majia pomelos which contained 50 g carbohydrate.This group of diabetic patients enrolled for the case control period.
Arm/Group | Diabetic | Healthy | Diabetic 2 - Without Pomelo | Diabetic 2 - With Pomelo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes